CLINICAL TRIAL: NCT01543191
Title: A Phase 1 Dose-escalation Study TO Evaluate the Safety and Tolerability of PUR118 and Placebo in Subjects With CF
Brief Title: A Safety and Tolerability Study OF PUR118 In Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 601-0009
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Cystic Fibrosis
Keywords: Lung Diseases; Respiratory Tract Diseases; Fibrosis
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases; Respiratory Tract Diseases; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PUR118 (Experimental)
  Interventions: Drug: PUR118
- Placebo (Placebo Comparator)
  Interventions: Drug: PUR118

INTERVENTIONS:
Drug: PUR118 — low dose and high dose for 3 doses, BID

SUMMARY:
The purpose of this study is to determine whether PUR118 is safe and tolerable in a population of subjects with Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-lactating healthy female.
* Age 18 to 55 years of age (inclusive) on day of signing informed consent.
* Subject has a BMI of 17 or greater.
* Subject has a confirmed diagnosis of cystic fibrosis documented by a compatible clinical or radiographic presentation, and definitive accepted lab and clinical criteria (e.g., sweat chloride > 60 mEq/L or 2 disease causing CFTR mutations) OR is regularly attending a Consultant led clinic where the diagnosis of Cystic Fibrosis is not in doubt.
* Subject has an FEV1 ≥ 45% of predicted at screening.
* Subject has an oxygen saturation >92% on room air as determined by pulse oximetry at screening.
* Subject is a non-smoker or ex-smoker has not smoked for at least six months prior to screening.
* Subject is otherwise medically stable without clinically significant abnormal screening results that depart from their usual baseline level of health as a subject with CF.
* Must be willing and able to communicate in English and participate in the whole study.
* Must provide written informed consent.

Exclusion Criteria:

* Subject has unstable lung disease, as defined by a change in medical regimen during the preceding 2-weeks, or a significant new finding on chest radiograph (pneumothorax, lobar/segmental collapse), or in the opinion of the Investigator, has had a decline in pulmonary status within the last year not considered a part of the usual, chronic progression of CF lung disease and part of their baseline health condition as a subject with CF.
* Subject has had an exacerbation of respiratory symptoms within the past 30 days that required initiation of a new or altered respiratory therapy.
* Subject had either an upper or lower respiratory illness within the 30 days prior to dosing days, or has symptoms from such an illness that have not resolved.
* Subject has a history of lung transplantation.
* Females of child bearing potential who are pregnant, or lactating. Females who are sexually active and either not surgically sterile or not willing to use an acceptable form of contraception
* Clinically significant abnormal biochemistry, haematology or urinalysis not consistent with CF as judged by the Investigator
* Failure to satisfy the Investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 4-6 weeks
  Changes in clinical signs and symptoms from physical examination and chest examination, changes in clinical safety laboratory tests, vital signs, spirometry, lung clearance index, 24-hour sputum weight and volume, oxygen saturation, ECG, telemetry, and adverse events.

SECONDARY OUTCOMES:
Pharmacodynamics | 36 hours
  To assess impact of PUR118 on mobilization and expectorated volume of airway mucus secretions.
  To evaluate impact of PUR118 on measurements of lung function, including ventilation inhomogeneity, by both spirometry and measurement of the lung clearance index (LCI).
  To evaluate an impact of PUR118 on sputum, serum and plasma biomarkers related to airway inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Smith, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Belfast, Northern Ireland, United Kingdom